CLINICAL TRIAL: NCT01068522
Title: Traumatic Brain Injury in Latin America: Lifespan Analysis
Brief Title: Study to Improve Outcomes for Survivors of Traumatic Brain Injury in Latin America
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33888-B; 1R01NS058302 (NIH)
Record Dates: First submitted 2010-02-11; First posted 2010-02-15 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Traumatic Brain Injury; Brain Injuries
Keywords: Intracranial pressure; Intracranial pressure monitoring; Head injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICP monitoring (Experimental): Care based upon intracranial pressure.
  Interventions: Device: Parenchymal Intracranial pressure monitor
- Usual Care (Active Comparator): Treatment based on clinical and imaging without intracranial pressure monitoring.
  Interventions: Other: Treatment based on clinical and imaging observations

INTERVENTIONS:
Device: Parenchymal Intracranial pressure monitor — Treatment based on readings from Parenchymal intracranial pressure monitor.
  Other Names: Integra Life Sciences Camino Intracranial Monitor
  Arms: ICP monitoring
Other: Treatment based on clinical and imaging observations — Treatment based on clinical and imaging observations.
  Arms: Usual Care

SUMMARY:
People who survive severe traumatic brain injury (TBI) live with profound cognitive impairments that alter their developmental course and define their future possibilities. Worldwide, TBI is the leading cause of death and disability among children and adolescents (Murgio, 2000). In the United States, the annual incidence of TBI is six times greater than that of multiple sclerosis, HIV/AIDS, spinal cord injury, and breast cancer combined [Centers for Disease Control, American Cancer Society, National Multiple Sclerosis Society]. The burden of TBI may be even greater in developing countries, due to civil unrest and war, and to the absence of mandated prevention such as seat belt laws.

The long-term objective of the investigators' research group is to improve outcomes for survivors of TBI in Latin America. To that end, the investigators have created a structure for professionals and institutions involved in the treatment of TBI to generate research; to facilitate education, standardization, certification, the dissemination of information and resources; and to foster the development of evidence-based guidelines. The structure is the Latin American Brain Injury Consortium (LABIC).

DETAILED DESCRIPTION:
The objective of this application is to establish a network of Centers of Excellence within LABIC that will, in collaboration with U.S. partners, conduct research and training programs about TBI. To that end, this project will include scientific investigation and capacity building.

The primary focus for scientific investigation is to conduct a high quality randomized controlled trial addressing a question of critical importance to the management of TBI worldwide:

• Does the use of information provided by intracranial pressure (ICP) monitoring to direct treatment of patients with TBI improve medical practice and patient outcomes in a developing country? This trial will be conducted in three trauma centers in Bolivia, in which the infrastructures and practice patterns are optimal for strong internal validity, while at the same time the level of resources is representative of trauma care as practiced in the developing world.

The secondary focus for scientific investigation is to conduct a prospective study of TBI in seven trauma centers in Bolivia, Brazil, Argentina, Colombia, and Ecuador that represent the variation in access to and use of resources in the developing world. This study will address two questions of vital importance to management of TBI in developing countries:

* To what extent do the findings from the randomized trial about ICP monitoring in particular, and brain injury care in general, generalize to diverse populations of TBI patients in Latin America?
* What is the association between resources and outcomes from TBI in developing countries? To build capacity, we will provide education, equipment, and structure, and will foster the collaborations established during the pilot R21 phase of this project. Our commitment is that LABIC becomes completely independent as a research entity. At the end of the funding period LABIC constituents will be able to identify important research questions, design the research, write successful proposals for funding, carry out strong studies, analyze and interpret the data, submit successful publications to internationally recognized peer reviewed journals, and disseminate information across Latin America.

Our specific aims are:

Specific Aim#1: In a randomized controlled trial in 3 trauma centers in Bolivia, test the effect on outcomes of management of severe TBI guided by information from ICP monitors vs. a standard empiric protocol.

Hypothesis #1: Patients with severe TBI whose acute care treatment is managed using ICP monitors will have significantly lower mortality and better neuropsychological and functional recovery at 6 months post-trauma than those whose treatment is managed with the standard protocol.

Hypothesis #2: The incorporation of ICP monitoring into the care of patients with severe TBI will minimize secondary complications and decrease length of stay in intensive care unit (ICU).

Specific Aim #2: In a prospective, observational study conducted in trauma centers in Latin America, test the association between resource availability/medical management and outcomes for patients with severe TBI.

Hypothesis #3: The association between treatment and outcomes for patients with severe TBI identified in the randomized trial of ICP monitoring will generalize to the population in the prospective, observational, multi-center, multi-national study.

Hypothesis #4: Variations in resource availability and medical management will be significantly associated with mortality and functional recovery for patients with severe TBI, after controlling for patient and injury characteristics.

Specific Aim #3: Establish a network of research centers with investigators trained and skilled in the design, conduct, and funding of research programs to address TBI and other brain disorders in Latin America.

In fulfilling these aims, we will answer important research questions about patient characteristics, treatment, and outcomes from TBI in an environment of limited resources, aspects of which will generalize to other developing countries as well as to the developed world. In a developing country, we will test the effectiveness of technology considered pivotal to brain trauma treatment in the developed world - the ICP monitor. The outcome of this trial may serve to standardize practice, improve outcomes, and mobilize resources worldwide. A randomized controlled trial of ICP monitoring has never been performed. As specifically stated in the Guidelines for the Management of Severe Brain Injury (Bullock et al., 1996), this is a critical gap in the evidence base that supports the role of ICP monitoring in TBI care. As such, the results of the RCT as performed in Bolivia will have global implications regardless of the level of development of the trauma system.

We will also establish sustainable capacity to conduct research about TBI in Latin America. Within the structure of LABIC, we will create a cadre of professionals who are trained in clinical research and equipped to carry out studies that answer questions important to Latin America. These studies will establish a literature base from which Latin American treatment guidelines will be generated. With training in cognitive assessment, we will introduce a new discipline into many of the Latin American medical systems that will provide an understanding of the unique and profound disabilities associated with brain disorders.

ELIGIBILITY:
Inclusion Criteria:

* admission to study hospital within 24 hours of injury
* closed head trauma
* Glasgow Coma Scale (GCS) < 8 on admission or if intubated, GCS Motor < 5, within first 48 hours after injury
* No foreign object in brain parenchyma
* Randomized:

  * within 24 hours of injury [for patients with GCS < 8 on admission] or
  * within 24 hours of deterioration [patients deteriorating to GCS < 8 within 48 hours of injury]
* Age > 12

Exclusion Criteria:

* GCS of 3 with bilateral fixed and dilated pupils and/or decision to not actively treat prior to enrolment into study
* No beds available in ICU
* No ICP monitor available
* Pregnancy
* Prisoner
* No consent
* Non-survivable injury
* Other (e.g., Pre-injury life expectancy under 1 year)
* Pre-existing neurological disability that would not allow follow-up

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
In a randomized controlled trial in 3 trauma centers in Bolivia, test the effect on outcomes of management of severe TBI guided by information from ICP monitors vs. a standard empiric protocol. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Randall M Chesnut, MD, Principal Investigator — University of Washington, Harborview Medical Center, Seattle, WA
Locations (6):
- Bolivia (4):
  - Hospital Viedma, Cochabamba
  - Hospital Japones, Santa Cruz de la Sierra
  - Hospital San Juan de Dios, Santa Cruz de la Sierra
  - Hospital San Juan de Dios, Tarija
- Ecuador (2):
  - Hospital de Especialidades Eugenio Espejo, El Ángel
  - Hospital Luis Vernaza, Guayaquil

REFERENCES:
- [Derived] Chesnut RM, Temkin N, Carney N, Dikmen S, Rondina C, Videtta W, Petroni G, Lujan S, Pridgeon J, Barber J, Machamer J, Chaddock K, Celix JM, Cherner M, Hendrix T; Global Neurotrauma Research Group. A trial of intracranial-pressure monitoring in traumatic brain injury. N Engl J Med. 2012 Dec 27;367(26):2471-81. doi: 10.1056/NEJMoa1207363. Epub 2012 Dec 12. PMID 23234472